CLINICAL TRIAL: NCT02707614
Title: Perioperative Mechanisms for Postoperative Function - the Case of Prostastectomy
Brief Title: Why in PACU After Prostastectomy 2016
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Dr, DMSci, Rigshospitalet, Denmark
Other Study IDs: PACU Prostastectomy 2016
Record Dates: First submitted 2016-03-01; First posted 2016-03-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Perioperative, Enhanced Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Robotic vs open prostastectomy: One group is operated by open prostatectomy the other by robotic assistance
  Interventions: Procedure: Robotic vs open prostastectomy

INTERVENTIONS:
Procedure: Robotic vs open prostastectomy — robotic minimal invasive surgery

SUMMARY:
This study aims to describe the postoperative functions of patients after undergoing open or robotic prostastectomy. Primary endpoints will focus on complications in the post-anaesthesia care unit (PACU) which prevent dischard from PACU to the general ward. This include Aldrete scores and other complications that can be registrered descriptively. Furthermore, the study seeks to compare what influence open versus robotic prostastectomy have on peri- og postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Histology diagnosis of prostate cancer
* Surgery intended for removal or staging of prostate cancer: open prostatectomy, robotic prostastectomy, open staging surgery, laparoscopic staging surgery.

Exclusion Criteria:

* Patients with prostate cancer that do not have surgery.
* Surgery regarding only removal of distant mestatases origined from prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes male patients with prostate cancer that will undergo surgery regarding removal or staging of their prostate cancer. The stage of the disease is insignificant, however the patients preoperative physical state for surgery will be registrered in detailed such as comorbidities, height, weight, bloodpressure and blood test results.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Complications | up to 7 days
  Complications assessed by aldrete score

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, abdominal center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided